CLINICAL TRIAL: NCT05103826
Title: A Phase I Study to Evaluate Safety 、Tolerability 、 Pharmacokinetics and Efficacy of SHR6390 in Combination With Famitinib in the Treatment of ER + / HER2- Advanced Breast Cancer
Brief Title: A Study of SHR6390 Combined With Famitinib in the Treatment of ER + / HER2- Advanced Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor R & D Strategy Adjustment
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR6390-SHR1020-I-101-BC
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: ER+ / HER2- Advanced Breast Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR6390+famitinib (Experimental): Participants will receive SHR6390 in combination with famitinib.
  Interventions: Drug: SHR6390、Famitinib

INTERVENTIONS:
Drug: SHR6390、Famitinib — SHR6390, oral;Famitinib, oral.

SUMMARY:
The study is being conducted to assess the safety 、tolerability 、 pharmacokinetics and efficacy of SHR6390 combined with famitinib in the treatment of ER + / HER2- advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects aged 18 to 75 years old；
2. ECOG performance status 0-1;
3. Life expectancy is not less than 12 weeks;
4. Histological or cytological confirmation of ER+/HER2- recurrent/metastatic breast cancer;
5. Participants with measurable disease must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST1.1;
6. Adequate function of major organs;
7. Voluntary participation in the study, signed informed consent, good compliance and willingness to cooperate with follow-up.

Exclusion Criteria:

1. Confirmed diagnosis of HER2 positive disease;
2. Participants who previously received SHR6390 or VEGFR inhibitors;
3. Allergy to study drug or its components;
4. Participated in other drug clinical trials within 4 weeks before the first dose;
5. Other malignancies within 3 years, except cured non-melanoma skin cancer , skin basal cell carcinoma and squamous-cell carcinoma or carcinoma in situ of the cervix;
6. Clinically significant cardiovascular and cerebrovascular diseases,including but not limited to severe acute myocardial infarction within 6 months before enrollment, unstable or severe angina, Congestive heart failure (New York heart association (NYHA) class > 2), or ventricular arrhythmia which need medical intervention；
7. Tumor has invaded important blood vessels or the tumor is likely to invade important blood vessels and cause fatal hemorrhage during treatment;
8. Urine routine test indicates urine protein ≥(++), or 24-hour urine protein >1.0g;
9. Active HBV/HCV/HIV infection;
10. The investigators determined that other conditions were inappropriate for participation in this clinical trial；
11. Pregnant or breast-feeding women;
12. Central nervous system (CNS) invasion.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
(Safety Lead-in) dose limited toxicity (DLT) of SHR6390+famitinib in the first cycle | up to 28 days
(Safety Lead-in) Recommended Phase II Dose (RP2D) of SHR6390+famitinib | up to 28 days

SECONDARY OUTCOMES:
AEs+SAEs | up to 24 months
  from the first drug administration to within 30 days for the last treatment dose
Evaluation of pharmacokinetic parameter of SHR6390+famitinib: Cmax | 6 months
Evaluation of pharmacokinetic parameter of SHR6390+famitinib: Tmax | 6 months
Evaluation of pharmacokinetic parameter of SHR6390+famitinib: t1/2 | 6 months
Evaluation of pharmacokinetic parameter of SHR6390+famitinib: AUC | 6 months
Evaluation of pharmacokinetic parameter of SHR6390+famitinib: CL/F | 6 months
Evaluation of pharmacokinetic parameter of SHR6390+famitinib: Vz/F | 6 months
Evaluation of pharmacokinetic parameter of SHR6390+famitinib: Rac | 6 months
Objective Response Rate (ORR) | up to 24 months
  Number of responders Assessed by Modified Response Evaluation Criteria In Solid Tumours (RECIST v1.1) for target lesions assessed by CT or MRI
Disease control rate (DCR) | up to 24 months
  Complete response + Partial response + Stable disease (CR+PR+SD) based on RECIST 1.1
Duration of response (DoR) | up to 24 months
  Time from documentation of tumor response to disease progression assessed among patients who had an objective response

CONTACTS AND LOCATIONS:
Locations (1):
- Harbin Medical University Cancer Hospital, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided